CLINICAL TRIAL: NCT00622089
Title: An Open Label Follow-On Study of Safety and Pharmacodynamic Effects of 24 Weeks of Treatment With DIO-902 in Combination With Metformin and Atorvastatin in Subjects With Type 2 Diabetes Mellitus (Protocol No. DIO-503)
Brief Title: Open Label Safety & Pharmacodynamic Study 24Wk w/DIO-902 Combo w/Metformin & Atorvastatin in T2DM Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Program terminated
Sponsor: DiObex (Industry)
Responsible Party: Bernice Welles, MD, DiObex, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIO-503
Record Dates: First submitted 2008-01-03; First posted 2008-02-22 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; type 2 diabetes; cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 150mg DIO-902 + 10mg Atorvastatin
  Interventions: Drug: DIO-902
- 2. (Experimental): 300mg DIO-902 + 10mg Atorvastatin
  Interventions: Drug: DIO-902
- 3 (Experimental): 450mg DIO-902 + 10mg Atorvastatin
  Interventions: Drug: DIO-902

INTERVENTIONS:
Drug: DIO-902 — 150mg DIO-902 + 10mg atorvastatin
  Arms: 1
Drug: DIO-902 — 300mg dose once per day for 24 weeks
  Arms: 2.
Drug: DIO-902 — 450mg dose once per day for 24 weeks
  Arms: 3

SUMMARY:
DiObex Inc. is developing an experimental drug (DIO-902) that is made up of part of the ketoconazole molecule for the treatment of elevated blood glucose associated with type 2 diabetes mellitus. Ketoconazole (Nizoral®) is a drug available by prescription for the treatment of fungal infections however DIO-902 is an investigational drug. DIO-902 may lower blood glucose by lowering levels of a naturally occurring hormone called cortisol. Elevated cortisol may contribute to the development of type 2 diabetes.

DETAILED DESCRIPTION:
To maintain the blind in Protocol DIO-502, subjects will be re-randomized at Study Visit 1 to one of three doses of DIO-902: 150, 300 or 450 mg QHS. All subjects receiving DIO-902 placebo and 50% of subjects receiving DIO-902 will be re-randomized to one of three DIO-902 doses. The remaining 50% of subjects receiving DIO-902 will be assigned to their original DIO-902 dose. The re- randomization will be performed by a group independent of study conduct to ensure the treatment status of the subject while in Protocol DIO-502 remains blinded. In addition, subjects will continue on the same dose of metformin that they had been taking during the conduct of Protocol DIO-502. Subjects will continue on atorvastatin 10 mg for the first 4 weeks of this protocol. Thereafter, at Study Visits 3 and 4, the dose of atorvastatin may be increased up to a maximum of 40 mg daily in order to achieve LDL-cholesterol/non-HDL cholesterol goals specified within the protocol. In addition, after Study Visit 4 (Week 12) subjects with HbA1c levels of > 7.5% (0.075 Hb Fract.) will undergo a one time titration of their oral hypoglycemic regimen as per the algorithm provided in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participated in DIO-502

Exclusion Criteria:

* Did not participate in DIO-502

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The following parameters will be evaluated at Week 12 and Week 24: • Proportion of subjects who reach the lipid goal as defined in the protocol from baseline • Proportion of subjects who meet the HbA1c goal as defined in the protocol from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United States (12):
  - Dr. Terence Hart, Muscle Shoals, Alabama
  - Genova Research, Tucson, Arizona
  - Research Solutions, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - Advanced Medical Research, Lakewood, California
  - Mills-Peninsula Helath Services, San Mateo, California
  - Diabetes Research Goup University of Hawaii at Manoa, Honolulu, Hawaii
  - Creighton Diabetes Center, Omaha, Nebraska
  - AHS Oklahoma Physician Group, Tulsa, Oklahoma
  - Covance Clinical Research Unit - Dr. Andrew Ahmann, Portland, Oregon
  - Covance CRU, Austin, Texas
  - Diabetes Glandular Disease Research Associates, San Antonio, Texas
- Australia (8):
  - Flinders Medical Centre, Adelaide, South Australia
  - Lyell McEwin Hospital, North Western Adelaide, South Australia
  - ECRU, Box Hill, Melbourne, Victoria
  - School of Medicine and Pharmacology, Fremantle, Western Australia
  - Keough Institute, Nedands, Western Australia
  - Endocrinology Research Unit, Herston Road
  - Endocrinology Department, St Leonards
  - Royal Melbourn Hospital, Victoria
- New Zealand (4):
  - Middlemore Hospital, Otahuhu, Auckland
  - Lipid and Diabetes Research, Christchurch
  - Waikaito Hospital, Hamilton
  - Diabetes Centre, Wellington